CLINICAL TRIAL: NCT00502918
Title: Feasibility Study -Clinical Feasibility of Computerized Labor Monitor (CLM) -Heart Application
Brief Title: Clinical Feasibility of Computerized Labor Monitor (CLM) -Heart Application (HA)
Status: Terminated | Type: Observational
Why Stopped: The study was terimnated - low rate of cases
Sponsor: Barnev Ltd (Other)
Responsible Party: Clinical Trial Manager, Barnev Ltd
Other Study IDs: TASMC-07-AM-279-CTIL
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2007-07

CONDITIONS: Obstetrics; Labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Device: CLM - HA Continuous Monitoring System Heart Application

INTERVENTIONS:
Device: CLM - HA Continuous Monitoring System Heart Application

SUMMARY:
The study is a feasibility study to check the possibility of tracking the heart rate of the fetus and to translate the outcome to the progress of the labor

DETAILED DESCRIPTION:
Every year, millions of babies are born worldwide. Yet, despite great advances in medical technology, the method used to obtain the most critical parameter in labor management - cervix dilatation, remains a vaginal (manual) examination. This vaginal examination, intended to estimate the dilatation of the cervix and the progress of the baby's head, is inaccurate, non-continuous and involves the risk of infection to both fetus and mother. It is also uncomfortable to the mother. The consequences of infections or delayed treatment may range from simple complications to irreversible damage. Early detection of abnormal patterns of labor progress could prevent complications and shorten the labor process and hospitalization, thereby saving both aggravation and cost.

To truly manage the labor process, a labor management system is required. Such a system is expected to provide the obstetrical staff with the flow of accurate, continuous, real-time information, such as cervix dilatation.

ELIGIBILITY:
Inclusion Criteria:

1. Laboring women refered to the maternity center in active labor (3cm dilatation and contraction)
2. Gestational age 37-42 weeks. (GA)
3. Single Fetus.
4. Subjects who understand, agreed and signed the informed consent form.

Exclusion Criteria:

1. Women with abnormal placentation (Placenta previa) -
2. Abnormal fetal presentation (Breech presentation).
3. Maternal History of HIV and/or blood transmitted Hepatitis and /or active genital Herpes.
4. Need for immediate delivery (cord prolapsed or suspected placental abruption)

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Laboring women reffered to the maternity center in active labor (3cm - 7 cm) dilataion and contraction
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2008-07 (Estimated); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Monitoring fetal heart movement | During labour

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Many, MD, Principal Investigator — Sackler School od Medicine , Tel Aviv University
Locations (1):
- Tel Aviv Soraski medical center, Tel Aviv, Israel